CLINICAL TRIAL: NCT02533180
Title: Evaluation of Donor Specific Immune Senescence and Exhaustion as Biomarkers of Operational Tolerance Following Liver Transplantation in Adults (ITN056ST)
Brief Title: Evaluation of Donor Specific Immune Senescence and Exhaustion as Biomarkers of Tolerance Post Liver Transplantation
Acronym: OPTIMAL
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network); PPD Development, LP (Industry); Rho Federal Systems Division, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN056ST
Record Dates: First submitted 2015-08-21; First posted 2015-08-26 (Estimated); Results first posted 2021-03-05 (Actual); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Liver Transplant; Liver Transplantation
Keywords: Liver allograft recipient; Immunosuppression withdrawal; Calcineurin inhibitor (CNI) based immunosuppression; Living Donor (of the Respective Liver Transplant Recipient)

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Immunosuppression withdrawal (ISW) (Other): Gradual immunosuppression withdrawal according to the protocol defined algorithm
  Interventions: Biological: Immunosuppression withdrawal

INTERVENTIONS:
Biological: Immunosuppression withdrawal — Participants will initiate calcineurin inhibitor (CNI) withdrawal after at least 3 weeks of stable liver function, as documented by liver function tests (direct bilirubin, alanine aminotransferase and gamma-glutamyl transferase) separated by at least 1 week in the 3 week period prior to withdrawal.
  CNI withdrawal will occur in eight 3 week intervals with each subsequent reduction based on liver function tests over the prior 3 week interval.
  Participants on CNI and prednisone will undergo withdrawal from the two therapies concurrently.
  If participants are weaned off the CNI successfully, they will initiate non-CNI withdrawal. The non-CNI withdrawal includes two dose reductions of approximately 50% over a 6 week period each, after which the drug will be discontinued.
  Other Names: ISW

SUMMARY:
The primary aim of this study is to determine whether a peripheral blood or graft lymphocyte phenotype of immune senescence or exhaustion is different between operationally tolerant and non-tolerant liver allograft recipients.

DETAILED DESCRIPTION:
People who have liver transplants must take anti-rejection medication (immunosuppression) for the rest of their lives. If they stop, their immune system may reject the transplanted liver. All anti-rejection medications have side effects. Because of the side effects of anti-rejection medications, an important goal of transplant research is to allow people to accept their transplanted organ without long term use of anti-rejection medications. This is called tolerance. In this study, participants who received a liver transplant will have their anti-rejection medication(s) gradually reduced over a period of time and then stopped. The study calls this 'immunosuppression withdrawal'.

The purpose of this research study is to see how many people will develop tolerance after immunosuppression withdrawal. The researchers also want to find out if there are blood or liver biopsy tests that can help transplant doctors in the future predict whether it is safe to decrease or stop anti-rejection medications in people who received a liver transplant.

ELIGIBILITY:
Inclusion Criteria:

Recipient participants must meet all of the following criteria to be eligible for this study:

1. At the time of screening:

   * 18 to 50 years old and more than 6 years post-transplant OR
   * Greater than 50 years old and more than 3 years post-transplant
2. Recipient of either deceased or living donor liver transplant. Recipients of living donor transplants must have a donor who is also willing to enroll
3. Recipient of single organ transplant only
4. Must have a screening liver biopsy that fulfills the following criteria based on the central pathology reading:

   * Portal inflammation and interface activity is preferably absent, but minimal to focal mild portal mononuclear inflammation may be present. Interface necro-inflammatory activity is absent or equivocal/minimal and, if present, involves a minority of portal tracts and not generally associated with fibrosis
   * Negative for perivenular inflammation
   * Lymphocytic bile duct damage, ductopenia, and biliary epithelial senescence changes are absent unless there is an alternative, non-immunological explanation (e.g. biliary strictures)
   * Fibrosis (if present) should be mild overall, and portal-to-portal bridging should not be more than rare. Perivenular and peri-sinusoidal fibrosis should not be more than mild according to the Banff criteria
   * Findings for obliterative or foam cell arteriopathy are negative
5. Liver function tests (Direct bilirubin, alanine aminotransferase (ALT)), less than twice the upper limit of normal (ULN). ULN values for liver function tests will be defined by ranges from Harrison's Principles of Internal Medicine, 18th edition
6. Receiving calcineurin inhibitor (CNI) based maintenance immunosuppression. Participants may also concurrently receive:

   * Low dose mycophenolate mofetil (MMF ≤ 1500 mg daily) or mycophenolic acid (≤ 1080 mg daily), OR
   * Prednisone ≤ 7.5 mg daily, or equivalent corticosteroid
7. Ability to sign informed consent

Living donor participants must meet all of the following criteria to be eligible for this study:

1. At the time of screening: ≥18 years old
2. Living donor of the liver allograft of an enrolled recipient participant
3. Ability to sign informed consent
4. Willingness to donate appropriate biologic samples

Exclusion Criteria:

Recipient participants who meet any of the following criteria will not be eligible for this study:

1. History of hepatitis C virus (HCV) infection (defined as a positive HCV antibody test)
2. Positive antigen-antibody immunoassay for human immunodeficiency virus, HIV-1/2
3. Serum positivity for HBV surface antigen or HBV-DNA
4. History of immune-mediated liver disease in which immunosuppression discontinuation is inadvisable (autoimmune hepatitis, primary sclerosing cholangitis, primary biliary cirrhosis)
5. Any medical condition associated with a likely need for systemic corticosteroid administration, e.g., reactive airways disease
6. Prospective baseline liver biopsy showing any of the following: (see recipient inclusion criteria #4)

   * acute rejection according to the Banff global assessment criteria
   * early or late chronic rejection according to the Banff global assessment criteria
   * inflammatory activity and/or fibrosis in excess of permissive criteria according to Banff 2012 criteria
   * any other histological findings that might make participation in the trial unsafe. Eligibility will be determined by the findings on the central biopsy reading
7. Rejection within the 52 weeks prior to screening
8. Estimated glomerular filtration rate (GFR) <40 ml/min as calculated by CKD-EPI method (to mitigate the risk of worsening renal failure should rejection occur and high level of CNI be required)
9. The need for chronic anti-coagulation that cannot be safely discontinued for a minimum of 1 week to safely perform a liver biopsy
10. Pregnant females and females of childbearing age who are not using an effective method of birth control
11. Current drug or alcohol dependency
12. Inability to comply with the study visit schedule and required assessments, including frequent liver function monitoring and protocol biopsies
13. Inability to comply with study directed treatment
14. Any medical condition that in the opinion of the principal investigator would interfere with safe completion of the trial
15. Participation in another interventional clinical trial within the 4 weeks prior to screening

Living donor participants who meet any of the following criteria will not be eligible for this study:

1. Any medical condition, such as anemia, coagulopathy, etc., that in the opinion of the principal investigator would interfere with safe participation in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-12-15 (Actual); Primary Completion 2020-02-10 (Actual); Study Completion 2022-07-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James F. Markmann, MD, PhD, Study Chair — Massachusetts General Hospital: Transplantation
Locations (7):
- United States (7):
  - University of California, San Francisco Medical Center, San Francisco, California
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Baylor University Medical Center at Dallas, Dallas, Texas

REFERENCES:
- [Derived] Sanchez-Fueyo A, Markmann JF. Immune Exhaustion and Transplantation. Am J Transplant. 2016 Jul;16(7):1953-7. doi: 10.1111/ajt.13702. Epub 2016 Feb 16. PMID 26729653
- See also: ITN OPTIMAL Study Website — http://optimalstudy.org/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) — https://www.niaid.nih.gov/about/dait
- See also: National Institute of Allergy and Infectious Diseases (NIAID) — https://www.niaid.nih.gov/
- See also: Immune Tolerance Network (ITN) — http://www.immunetolerance.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 100 participants were enrolled from 7 sites in the US between December 2015 and November 2018. 61 of the enrolled participants were eligible to initiate immunosuppression withdrawal and the remaining 39 participants were terminated (e.g., ineligible to initiate immunosuppression withdrawal) based on biopsy findings or other pre-specified criteria.
Pre-assignment Details: Informed consent was obtained from potentially eligible individuals who then underwent a study-mandated biopsy to determine if they were allowed to initiate immunosuppression withdrawal based on pre-specified histological criteria.
Groups:
- Enrolled, Did Not Initiate Immunosuppression Withdrawal: Theses participants were consented and enrolled into the study, but did not initiate immunosuppression withdrawal as specified by the protocol.
- Initiated Immunosuppression Withdrawal: These participants were enrolled into the study and initiated immunosuppression withdrawal per protocol. Participants could initiate withdrawal from calcineurin inhibitor (CNI) monotherapy or combination therapy with CNI and prednisone or CNI and a mycophenolate compound. Immunosuppression withdrawal followed a pre-specified process with the goal of achieving complete discontinuation of all immunosuppressive medication between 24 and 45 weeks after initiation of withdrawal.
Period: Overall Study
Arm/Group | Enrolled, Did Not Initiate Immunosuppression Withdrawal | Initiated Immunosuppression Withdrawal
Started | 39 | 61
Completed | 0 | 50
Not Completed | 39 | 11
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 0 | 1
Not completed — Withdrawal by Subject | 2 | 5
Not completed — Screen Failure | 37 | 0
Not completed — Protocol Deviation | 0 | 1
Not completed — Non-compliance | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Enrolled, Did Not Initiate Immunosuppression Withdrawal | Initiated Immunosuppression Withdrawal | Total
Number analyzed (Participants) | 39 | 61 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 31 | 37 | 68
  >=65 years | 8 | 24 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (15.88) | 60.3 (12.07) | 56.7 (14.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 24 | 43 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 4 | 6
  Not Hispanic or Latino | 36 | 49 | 85
  Unknown or Not Reported | 1 | 8 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 6 | 7
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 2 | 0 | 2
  White | 33 | 50 | 83
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 2 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 39 | 61 | 100
Alanine Transaminase (ALT) [Mean (Standard Deviation); unit: U/L] — The average of two ALT results taken at screening and 7 (+/- 2 days) before initiation of immunosuppression withdrawal. Only participants that initiated immunosuppression withdrawal will have both measurements.
  Reference: A liver function test -Normal Value: 7- 41 U/L. Population: Only participants that initiated immunosuppression withdrawal will have both measurements.
  U/L
    number analyzed (Participants) | 0 | 61 | 61
    (all) |  | 23.8 (10.7) | 23.8 (10.7)
Gamma-glutamyl Transferase (GGT) [Mean (Standard Deviation); unit: U/L] — The average of two GGT results taken at screening and 7 (+/- 2 days) before initiation of immunosuppression withdrawal. Only participants that initiated immunosuppression withdrawal will have both measurements.
  Reference: A liver function test- Normal Value: 9 - 58 U/L Population: Only participants that initiated immunosuppression withdrawal will have both measurements.
  U/L
    number analyzed (Participants) | 0 | 61 | 61
    (all) |  | 34.2 (24.58) | 34.2 (24.58)
Time from transplant (years) [Mean (Standard Deviation); unit: Years] — The time from transplant to study enrollment in years.
  Years | 11.5 (7.99) | 9.1 (5.65) | 10.0 (6.73)
Estimated Glomerular filtration rate (eGFR) [Mean (Standard Deviation); unit: mL/min/1.73 m2] — The value collected immediately prior to the initiation of immunosuppression (IS) withdrawal. Only subjects that initiated IS withdrawal will have this measurement (unit of measure of mL/min/1.73m2). eGFR was estimated using the CKD-EPI Creatine Equation (2021). eGFR is a measure of kidney function & helps determine disease stage. A value < 15 indicates kidney failure, 15-29 severe loss of kidney function, 30-44 moderate to severe loss of kidney function, 45-59 mild to moderate loss of kidney function, 60-89 mild loss of kidney function, and 90+ indicates normal kidney function. Population: Only subjects that initiated immunosuppression withdrawal will have this measurement.
  mL/min/1.73 m2
    number analyzed (Participants) | 0 | 61 | 61
    (all) |  | 73.9 (17.66) | 73.9 (17.66)
Fibrosis Score (ISHAK) [Number; unit: Percent of participants] — The value collected on the baseline biopsy prior to the initiation of immunosuppression withdrawal. Only subjects that initiated immunosuppression withdrawal will have this measurement. The ISHAK score is a measurement of fibrosis (scarring of tissue) in the liver. This scale ranges from 0 to 6, with a higher score indicating more severe fibrosis. Population: Only subjects that initiated immunosuppression withdrawal will have this measurement.
  Percent of participants
    0: number analyzed (Participants) | 0 | 61 | 61
    0 |  | 49.2 | 49.2
    1: number analyzed (Participants) | 0 | 61 | 61
    1 |  | 44.3 | 44.3
    2: number analyzed (Participants) | 0 | 61 | 61
    2 |  | 6.6 | 6.6
Liver Allograft Function Score (LAFSc) [Number; unit: Percent of participants] — The value collected on the baseline biopsy prior to the initiation of immunosuppression withdrawal. Only subjects that initiated immunosuppression withdrawal will have this measurement. The LAFSc score is a measurement of fibrosis (scarring of tissue) in the liver. This scale ranges from 0 to 6, with a higher score indicating more severe fibrosis Population: Only subjects that initiated immunosuppression withdrawal will have this measurement.
  Percent of participants
    0: number analyzed (Participants) | 0 | 61 | 61
    0 |  | 27.9 | 27.9
    1: number analyzed (Participants) | 0 | 61 | 61
    1 |  | 34.4 | 34.4
    2: number analyzed (Participants) | 0 | 61 | 61
    2 |  | 19.7 | 19.7
    3: number analyzed (Participants) | 0 | 61 | 61
    3 |  | 13.1 | 13.1
    4: number analyzed (Participants) | 0 | 61 | 61
    4 |  | 4.9 | 4.9
NIDDK Liver Transplantation Database Quality of Life [Mean (Standard Deviation); unit: NIDDK QOL Score] — The value collected prior to the initiation of immunosuppression withdrawal (ISW). Only subjects that initiated ISW have this measurement. This is a patient-reported survey of health and is summarized into five domains-measures of disease (0-21 with higher score indicating worse quality), psychological status (0-5 with higher score indicating worse quality), personal function (0-4 with higher score indicating better quality), social and role function (0-20 with higher score indicating worse quality), and general health perception (0-10 with higher score indicating better quality). Population: Only subjects that initiated immunosuppression withdrawal will have this measurement
  NIDDK QOL Score
    Measures of disease domain: number analyzed (Participants) | 0 | 61 | 61
    Measures of disease domain |  | 7.4 (4.57) | 7.4 (4.57)
    Psychological status domain: number analyzed (Participants) | 0 | 61 | 61
    Psychological status domain |  | 2.1 (1.68) | 2.1 (1.68)
    Personal function domain: number analyzed (Participants) | 0 | 61 | 61
    Personal function domain |  | 2.6 (1.37) | 2.6 (1.37)
    Social and role function domain: number analyzed (Participants) | 0 | 61 | 61
    Social and role function domain |  | 4.1 (3.00) | 4.1 (3.00)
    General health perception domain: number analyzed (Participants) | 0 | 61 | 61
    General health perception domain |  | 8.1 (1.48) | 8.1 (1.48)
SF-36 [Mean (Standard Deviation); unit: SF-36 Component Score] — The value collected immediately prior to the initiation of immunosuppression withdrawal. Only subjects that initiated immunosuppression withdrawal will have this measurement. The 36-Item Short Form Survey (SF-36) is a patient-reported questionnaire to measure quality of life. There are eight different scales that can be summarized into two summary scores-Mental Component Score (MCS) and Physical Component Score (PCS). Each score ranges from 0-100, with a higher score indicating a better quality of life. Population: Only subjects that initiated immunosuppression withdrawal will have this measurement.
  SF-36 Component Score
    PCS: number analyzed (Participants) | 0 | 61 | 61
    PCS |  | 49.5 (9.05) | 49.5 (9.05)
    MCS: number analyzed (Participants) | 0 | 61 | 61
    MCS |  | 53.8 (8.14) | 53.8 (8.14)

OUTCOME MEASURES:

1. Primary Outcome: The Percent of Participants Who Achieve Operational Tolerance 52 Weeks After Completion of Immunosuppression Withdrawal.
Description: Participants are considered as successfully withdrawn from immunosuppression if they remain off immunosuppression for at least 52 weeks without evidence of rejection since enrollment and have a liver biopsy at 52 weeks following completion of immunosuppression withdrawal demonstrating histological stability and the absence of rejection per Banff global assessment criteria. This biopsy is assessed by the central pathologist. All participants who fail to complete immunosuppression withdrawal, regardless of reason, or fail to have a biopsy 52 weeks after completion of immunosuppression withdrawal will be considered to have failed.
Time Frame: From initiation of immunosuppression withdrawal through 52 weeks after stopping all immunosuppression
Population: Participants who initiated immunosuppression withdrawal
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Groups:
- Immunosuppression Withdrawal (ISW): These participants were enrolled into the study and initiated immunosuppression withdrawal per protocol. Participants could initiate withdrawal from calcineurin inhibitor (CNI) monotherapy or combination therapy with CNI and prednisone or CNI and a mycophenolate compound. Immunosuppression withdrawal followed a pre-specified process with the goal of achieving complete discontinuation of all immunosuppressive medication between 24 and 45 weeks after initiation of withdrawal.
Arm/Group | Immunosuppression Withdrawal (ISW)
Number analyzed (Participants) | 61
Percent of Participants | 16.4 [8.15 to 28.1]

2. Secondary Outcome: Proportion of Participants Who Develop Donor-Specific AlloAbs (DSA) or de Novo Anti-human Leukocyte Antigen Human Leukocyte Antigen (HLA) Antibodies
Description: HLA is a molecule formed by a complex of genes which encode cell-surface proteins responsible for the regulation of the immune system. This molecule is unique for each individual. HLA molecules are present in all cells and are responsible for helping the immune system distinguish between your own cells and foreign cells (like pathogens). However, when our immune system encounters HLA molecules from another individual (like during pregnancy, after blood transfusions or transplantation) it recognizes this as foreign and can generate anti-HLA antibodies. These anti-HLA antibodies could cause harm to the transplanted organ by recognizing its cells as foreign triggering the immune system to attack. This endpoint looks at the development of newly developed donor-specific antibodies (DSA). DSA are a subset of anti-HLA antibodies that are specific against the donor organ. These anti-HLA antibodies are categorized into two classes-class I and class II. The data shown is only for class II DSA.
Time Frame: From initiation of immunosuppression withdrawal to study completion, up to 4.5 years.
Population: Initiated immunosuppression withdrawal and have analyzable blood samples prior to and after initiating withdrawal
Measure: Number (95% Confidence Interval); unit: Percent of participants
Groups:
- Immunosuppression Withdrawal (ISW): Initiated immunosuppression withdrawal and have analyzable blood samples prior to and after initiating withdrawal
Arm/Group | Immunosuppression Withdrawal (ISW)
Number analyzed (Participants) | 52
Percent of participants | 26.9 [15.57 to 41.02]

3. Secondary Outcome: The Incidence of Acute Rejection, Steroid Resistant Rejection, and Chronic Rejection
Description: Incidence will be measured as the proportion of participants who have acute rejection (per Banff criteria), steroid resistant rejection (rejection requiring antibody treatment), and chronic rejection (per Banff criteria), separately. The endpoint is summarized with a two-sided, 95% exact binomial confidence interval.
Time Frame: From initiation of immunosuppression withdrawal to study completion, up to 4.5 years.
Population: Participants who initiated immunosuppression withdrawal
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Immunosuppression Withdrawal (ISW)
Number analyzed (Participants) | 61
Percent of participants
  Acute Rejection | 47.5 [34.60 to 60.73]
  Steroid Resistant Rejection | 0 [0 to 5.87]
  Chronic Rejection | 0 [0 to 5.87]

4. Secondary Outcome: The Severity of Acute Rejection, Steroid Resistant Rejection, and Chronic Rejection
Description: Severity is based on the Banff global assessment grade according to the central pathology reading of the liver biopsy. For an individual subject, the worst severity is reported. Acute rejection is categorized into mild (rejection infiltrate in a minority of triads that is generally mild and confined within the portal spaces), moderate (rejection infiltrate expanding most or all of the triads), or severe (rejection infiltrate expanding most or all of the triads with spillover into periportal areas and moderate to severe perivenular inflammation that extends into the hepatic parenchyma and is associated with perivenular hepatocyte necrosis). Chronic rejection is categorized into early (bile duct atrophy/loss and foam cell obliterative arteriopathy in <50% of the portal tracts) or late (early criteria but >50% of the portal tracts) stage. Steroid resistant rejection is always considered severe. The endpoint is summarized with a two-sided, 95% exact binomial confidence interval.
Time Frame: From initiation of immunosuppression withdrawal to study completion, up to 4.5 years.
Population: Participants who had acute, steroid-resistant, or chronic rejection.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Groups:
- Participants With Rejection: Participants who had acute, steroid-resistant, or chronic rejection.
Arm/Group | Participants With Rejection
Number analyzed (Participants) | 29
Percent of participants
  Acute Rejection, Mild | 75.9 [56.46 to 89.70]
  Acute Rejection, Moderate | 20.7 [7.99 to 39.72]
  Acute Rejection, Severe | 3.5 [0.09 to 17.76]
  Chronic Rejection, Early Stage | 0 [0 to 11.94]
  Chronic Rejection, Late Stage | 0 [0 to 11.94]
  Steroid Resistant Rejection | 0 [0 to 11.94]

5. Secondary Outcome: The Timing of Acute Rejection, Steroid Resistant Rejection, and Chronic Rejection
Description: Time is measured as the time (in days) from the initiation of immunosuppression withdrawal to the time of the first biopsy showing rejection (per Banff criteria).
Time Frame: From initiation of immunosuppression withdrawal to study completion, up to 4.5 years.
Population: Participants who had acute, steroid-resistant, or chronic rejection.Time to event data could not be reported as no events were observed for Chronic Rejection and Steroid Resistant Rejection
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Participants With Rejection
Number analyzed (Participants) | 29
Days
  The Timing of Acute Rejection | 232 (134.5)
  The Timing of Chronic Rejection: number analyzed (Participants) | 0
  The Timing of Steroid Resistant Rejection: number analyzed (Participants) | 0

6. Secondary Outcome: The Incidence of Graft Fibrosis in Tolerant Versus Non- Tolerant Patients.
Description: Fibrosis of the liver is the formation of an excessive accumulation of scar tissue in the liver. Graft fibrosis was measured two ways by the ISHAK scale and by Liver Allograft Fibrosis Score (LAFSc) via a liver biopsy. Both scales range from 0 to 6, with a higher score indicating more severe fibrosis. A subject is considered as having graft fibrosis if the score is greater than or equal to 2 at their last available biopsy after the initiation of immunosuppression withdrawal.
Time Frame: From initiation of immunosuppression withdrawal to study completion, up to 4.5 years.
Population: Participants who initiated immunosuppression withdrawal and have a biopsy available after the initiation of immunosuppression withdrawal.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Groups:
- Initiated Immunosuppression Withdrawal With Available Biopsy (Tolerant): Participants who initiated immunosuppression withdrawal and have a biopsy available after the initiation of immunosuppression withdrawal and deemed tolerant by the primary endpoint.
- Initiated Immunosuppression Withdrawal With Available Biopsy (Non-tolerant): Participants who initiated immunosuppression withdrawal and have a biopsy available after the initiation of immunosuppression withdrawal and deemed non-tolerant by the primary endpoint.
Arm/Group | Initiated Immunosuppression Withdrawal With Available Biopsy (Tolerant) | Initiated Immunosuppression Withdrawal With Available Biopsy (Non-tolerant)
Number analyzed (Participants) | 10 | 41
Percent of participants
  ISHAK | 0 [0 to 30.85] | 12.2 [4.08 to 26.20]
  Liver Allograft Fibrosis Score | 50.0 [18.71 to 81.29] | 48.8 [32.88 to 64.87]

7. Secondary Outcome: The Progression of Graft Fibrosis in Tolerant Versus Non- Tolerant Patients
Description: Fibrosis of the liver is the formation of an excessive accumulation of scar tissue in the liver. Graft fibrosis was measured two ways by the ISHAK scale and by Liver Allograft Fibrosis Score (LAFSc) via a liver biopsy. Both scales range from 0 to 6, with a higher score indicating more severe fibrosis. Progression was calculated as the final available biopsy score minus the baseline biopsy score. A positive value indicates a worsening of fibrosis.
Time Frame: From initiation of immunosuppression withdrawal to study completion, up to 4.5 years.
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Fibrosis Score
Arm/Group | Initiated Immunosuppression Withdrawal With Available Biopsy (Tolerant) | Initiated Immunosuppression Withdrawal With Available Biopsy (Non-tolerant)
Number analyzed (Participants) | 10 | 41
Fibrosis Score
  ISHAK | 0 (0.94) | 0.2 (0.79)
  Liver Allograft Fibrosis Score | 0.1 (1.73) | 0.3 (1.44)

8. Secondary Outcome: The Incidence of Graft Loss
Description: A participant is considered to have graft loss when the donated liver needs to be removed and the participant is retransplanted with another donor liver or the participant is listed for retransplant. The endpoint will be summarized with a two-sided, 95% exact binomial confidence interval.
Time Frame: From initiation of immunosuppression withdrawal to study completion, up to 4.5 years.
Population: Participants who initiated immunosuppression withdrawal
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Immunosuppression Withdrawal (ISW)
Number analyzed (Participants) | 61
Percent of participants | 0 [0 to 5.87]

9. Secondary Outcome: The Incidence of All-Cause Mortality
Description: This number reflects all deaths observed in all participants in the study period, regardless of the cause. The endpoint will be summarized with a two-sided, 95% exact binomial confidence interval.
Time Frame: From initiation of immunosuppression withdrawal to study completion, up to 4.5 years.
Population: Participants who initiated immunosuppression withdrawal
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Immunosuppression Withdrawal (ISW)
Number analyzed (Participants) | 61
Percent of participants | 3.3 [0.40 to 11.35]

10. Secondary Outcome: The Incidence of Study-related SAEs
Description: An adverse event is considered a serious adverse event (SAE) if it results it any one of the following: death, life-threatening, inpatient hospitalization or prolongation of existing hospitalization, persistent or significant incapacity or substation disruption to conduct normal life functions, congenital anomaly or birth defect, or an important medical event. The event is considered study related if the medical monitor deems it to be at least possibly or definitely related to any of the study interventions/procedures (immunosuppression withdrawal, the blood draw, or the liver biopsy). The endpoint will be summarized with a two-sided, 95% exact binomial confidence interval.
Time Frame: From initiation of immunosuppression withdrawal to study completion, up to 4.5 years.
Population: Participants who initiated immunosuppression withdrawal
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Immunosuppression Withdrawal (ISW)
Number analyzed (Participants) | 61
Percent of participants | 16.4 [8.15 to 28.09]

11. Secondary Outcome: The Proportion of Operationally Tolerant Subjects Who Remain Free of Rejection at 3 Years After Completing Immunosuppression Withdrawal.
Description: Participants are considered operationally tolerant if they remain off immunosuppression for at least 52 weeks without evidence of rejection since enrollment and have a liver biopsy at 52 weeks following completion of immunosuppression withdrawal demonstrating histological stability and the absence of rejection per Banff global assessment criteria (as assessed by the central pathologist). This number reflects the participants that continue to show the absence of rejection per the Banff global assessment criteria (as assessed by the central pathologist) in the 3 years following completion of immunosuppression withdrawal. The endpoint will be summarized with a two-sided, 95% exact binomial confidence interval.
Time Frame: From initiation of immunosuppression withdrawal through 3 years after completing immunosuppression withdrawal.
Population: Participants who achieved operational tolerance as defined by the primary endpoint.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Groups:
- Operationally Tolerant: Participants who achieved operational tolerance as defined by the primary endpoint.
Arm/Group | Operationally Tolerant
Number analyzed (Participants) | 10
Percent of participants | 100 [69.15 to 100]

12. Secondary Outcome: Changes in Renal Function (Defined as Estimated GFR Calculated by the CKD-EPI Creatine Equation 2021) in Tolerant Versus Non-tolerant Participants at 1, 2 and 3 Years After Completing Immunosuppression Withdrawal.
Description: Glomerular filtration rate (GFR) is a measure of kidney function and helps determine the stage of kidney disease. A value less than 15 indicates kidney failure, 15 to 29 indicates severe loss of kidney function, 30 to 44 indicates moderate to severe loss of kidney function, 45 to 59 mild to moderate loss of kidney function, 60 to 89 indicates mild loss of kidney function, and 90 or higher indicates normal kidney function. The equation developed by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) is used to estimate GFR from serum creatinine. The baseline value was selected as the value collected immediately prior to the initiation of immunosuppression withdrawal. The year 1, 2, and 3, values are the values closest to and within 2 months of the expected date. Change was calculated as the year 1, 2, or 3 value minus baseline. A positive value indicates an increase in kidney function.
Time Frame: From initiation of immunosuppression withdrawal to study completion, up to 4.5 years.
Population: Participants who initiated immunosuppression withdrawal
Measure: Mean (Standard Deviation); unit: ml/min/1.73 m^2
Groups:
- Initiated Immunosuppression Withdrawal (Tolerant): Participants who initiated immunosuppression withdrawal and were deemed tolerant by the primary endpoint.
- Initiated Immunosuppression Withdrawal (Non-tolerant): Participants who initiated immunosuppression withdrawal and were deemed non-tolerant by the primary endpoint.
Arm/Group | Initiated Immunosuppression Withdrawal (Tolerant) | Initiated Immunosuppression Withdrawal (Non-tolerant)
Number analyzed (Participants) | 10 | 51
ml/min/1.73 m^2
  1 Yeaar | 4.8 (13.67) | 0 (13.85)
  2 Years | 4.2 (21.32) | -4.0 (12.19)
  3 year | -2.8 (18.11) | -2.6 (13.85)

13. Secondary Outcome: Changes in Quality of Life in Tolerant Versus Non-tolerant Participants and in All Participants at Baseline Versus the End of Study Participation, as Measured by the NIDDK Liver Transplantation Database Quality of Life Form.
Description: NIDDK Liver Transplantation Database Quality of Life Form is a patient-reported survey of patient health. The questionnaire is summarized into five domains-measures of disease (ranges from 0-21 with higher score indicating worse quality), psychological status (ranges from 0-5 with higher score indicating worse quality), personal function (ranges from 0-4 with higher score indicating better quality), social and role function (ranges from 0 to 20 with higher score indicating worse quality), and general health perception (ranges from 0 to 10 with higher score indicating better quality). Change was calculated as the difference between the questionnaire completed at the initiation of withdrawal and the questionnaire completed closest to the end of study participation. This change was calculated separately for tolerant and non-tolerant subjects.
Time Frame: From initiation of immunosuppression withdrawal to study completion, up to 4.5 years.
Population: Participants who initiated immunosuppression withdrawal and completed a NIDDK Liver Transplantation Database Quality of Life survey at baseline and after immunosuppression withdrawal initiation.
Measure: Mean (Standard Deviation); unit: Domain Score
Arm/Group | Initiated Immunosuppression Withdrawal (Tolerant) | Initiated Immunosuppression Withdrawal (Non-tolerant)
Number analyzed (Participants) | 9 | 47
Domain Score
  Measures of disease domain | -1.9 (5.69) | 0.5 (4.31)
  Psychological status domain | -0.6 (2.07) | 0.2 (1.43)
  Personal function domain | 0.1 (1.73) | -0.2 (1.14)
  Social and role function domain | 1.7 (2.89) | 1.1 (2.92)
  General health perception domain | -0.8 (2.11) | -0.5 (2.03)

14. Secondary Outcome: Changes in SF-36 in Tolerant Versus Non-tolerant Participants and in All Participants at Baseline Versus the End of Study Participation.
Description: SF-36 is a patient-reported survey of patient health. There are eight different scales that can be summarized into two summary scores-Mental Component Score and Physical Component Score. Each score ranges from 0-100, with a higher score indicating a better quality of life. Change was calculated as the difference between the questionnaire completed at the initiation of withdrawal and the questionnaire completed closest to the end of study participation. This change was calculated separately for tolerant and non-tolerant subjects.
Time Frame: From initiation of immunosuppression withdrawal to study completion, up to 4.5 years.
Population: Participants who initiated immunosuppression withdrawal and completed a SF-36 survey at baseline and after immunosuppression withdrawal initiation.
Measure: Mean (Standard Deviation); unit: SF-36 Component Score
Arm/Group | Initiated Immunosuppression Withdrawal (Tolerant) | Initiated Immunosuppression Withdrawal (Non-tolerant)
Number analyzed (Participants) | 9 | 45
SF-36 Component Score
  Physical Component Score | -3.4 (8.75) | -1.9 (7.72)
  Mental Component Score | 0.5 (9.75) | -0.7 (7.45)

15. Secondary Outcome: Predictive Value of the Following Parameters With Regard to Operational Tolerance: Time Post-transplant.
Description: Time post-transplant is calculated as time in years from transplant to enrollment. Participants are considered operationally tolerant if they remain off immunosuppression for at least 52 weeks without evidence of rejection since enrollment and have a liver biopsy at 52 weeks following completion of immunosuppression withdrawal demonstrating histological stability and the absence of rejection per Banff global assessment criteria (as assessed by the central pathologist). The odds ratio and corresponding 95% confidence interval are presented. The odds ratio represents the probability of achieving operational tolerance per year increase in time post-transplant. An odds ratio greater than 1 means that as the factor increases, operational tolerance is more likely to occur. Whereas less than 1 means operational tolerance is less likely to occur. Since the confidence interval contains 1, this means that as the corresponding factor increases, the likelihood of tolerance does not change.
Time Frame: From initiation of immunosuppression withdrawal to study completion, up to 4.5 years.
Population: Participants who initiated immunosuppression withdrawal
Measure: Number (95% Confidence Interval); unit: Probability of operational tolerance
Arm/Group | Immunosuppression Withdrawal (ISW)
Number analyzed (Participants) | 61
Probability of operational tolerance | 0.994 [0.864 to 1.144]

16. Secondary Outcome: Predictive Value and the Correlative Value of the Following Parameters With Regard to Operational Tolerance: Recipient Age.
Description: Recipient age is the age at the time of enrollment. Participants are considered operationally tolerant if they remain off immunosuppression for at least 52 weeks without evidence of rejection since enrollment and have a liver biopsy at 52 weeks following completion of immunosuppression withdrawal demonstrating histological stability and the absence of rejection per Banff global assessment criteria (as assessed by the central pathologist). The odds ratio and corresponding 95% confidence interval are presented. The odds ratio represents the probability of achieving operational tolerance per year increase in recipient age. An odds ratio greater than 1 means that as the factor increases, operational tolerance is more likely to occur. Whereas less than 1 means operational tolerance is less likely to occur. Since the confidence interval contains 1, this means that as the corresponding factor increases, the likelihood of tolerance does not change.
Time Frame: From initiation of immunosuppression withdrawal to study completion, up to 4.5 years.
Population: Participants who initiated immunosuppression withdrawal
Measure: Number (95% Confidence Interval); unit: Probability of operational tolerance
Arm/Group | Immunosuppression Withdrawal (ISW)
Number analyzed (Participants) | 61
Probability of operational tolerance | 0.982 [0.922 to 1.045]

ADVERSE EVENTS:
Time Frame: Up to 4.5 years
Description: Prior to initiating immunosuppression withdrawal, only adverse events and serious adverse events associated with protocol-mandated blood draws or the screening biopsy will be collected from study enrollment until initiation of immunosuppression withdrawal.
Arm/Group | Enrolled, Did Not Initiate Immunosuppression Withdrawal | Initiated Immunosuppression Withdrawal
All-Cause Mortality (participants affected / at risk) | 0/39 | 2/61
Serious Adverse Events (participants affected / at risk) | 0/39 | 27/61
Other Adverse Events (participants affected / at risk) | 3/39 | 53/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled, Did Not Initiate Immunosuppression Withdrawal (N=39) | Initiated Immunosuppression Withdrawal (N=61)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0)
Arrhythmia (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0)
Parotid gland enlargement (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 3 (7)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0)
Incarcerated hernia (General disorders) | 0 (0) | 0 (0)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 1 (2)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Haemobilia (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic artery stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0)
Intrahepatic portal hepatic venous fistula (Hepatobiliary disorders) | 0 (0) | 1 (1)
Transplant rejection (Immune system disorders) | 0 (0) | 5 (6)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 1 (1)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 3 (3)
Chlamydial infection (Infections and infestations) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0)
Hepatitis B (Infections and infestations) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 1 (1)
Lyme disease (Infections and infestations) | 0 (0) | 0 (0)
Medical device site joint infection (Infections and infestations) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0)
Post procedural cellulitis (Infections and infestations) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (3)
Viral infection (Infections and infestations) | 0 (0) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Transplant dysfunction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 0 (0)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 0 (0)
Laboratory test abnormal (Investigations) | 0 (0) | 0 (0)
Liver function test abnormal (Investigations) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 1 (1)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1)
Chest Pain (General disorders) | 0 (0) | 1 (1)
Corona virus infection (Infections and infestations) | 0 (0) | 1 (1)
Extremity necrosis (Vascular disorders) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Ageusia (Nervous system disorders) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 (0) | 0 (0)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Enrolled, Did Not Initiate Immunosuppression Withdrawal (N=39) | Initiated Immunosuppression Withdrawal (N=61)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Haemolytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Normochromic normocytic anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 2 (2)
Atrioventricular block (Cardiac disorders) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 3 (3)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0)
Intestinal ischaemia (Gastrointestinal disorders) | 0 (0) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Parotid gland enlargement (Gastrointestinal disorders) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gait disturbance (General disorders) | 0 (0) | 1 (1)
Incarcerated hernia (General disorders) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0)
Haemobilia (Hepatobiliary disorders) | 0 (0) | 0 (0)
Hepatic artery stenosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 1 (1)
Intrahepatic portal hepatic venous fistula (Hepatobiliary disorders) | 0 (0) | 0 (0)
Transplant rejection (Immune system disorders) | 0 (0) | 28 (28)
Abdominal wall abscess (Infections and infestations) | 0 (0) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 2 (2)
Bronchitis (Infections and infestations) | 0 (0) | 3 (4)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1)
Chlamydial infection (Infections and infestations) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 3 (3)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis norovirus (Infections and infestations) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 1 (1)
Hepatitis B (Infections and infestations) | 0 (0) | 1 (1)
Herpes virus infection (Infections and infestations) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 2 (2)
Influenza (Infections and infestations) | 0 (0) | 0 (0)
Lyme disease (Infections and infestations) | 0 (0) | 1 (1)
Medical device site joint infection (Infections and infestations) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Post procedural cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 4 (4)
Tooth infection (Infections and infestations) | 0 (0) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 6 (6)
Urinary tract infection (Infections and infestations) | 0 (0) | 5 (6)
Viral infection (Infections and infestations) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Arthropod bite (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Exposure to toxic agent (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Incisional hernia (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Meniscus injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural discomfort (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Synovial rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Transplant dysfunction (Injury, poisoning and procedural complications) | 0 (0) | 5 (6)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Blood glucose increased (Investigations) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 1 (1) | 5 (5)
Hepatic enzyme increased (Investigations) | 0 (0) | 2 (2)
Laboratory test abnormal (Investigations) | 0 (0) | 1 (1)
Liver function test abnormal (Investigations) | 0 (0) | 5 (5)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0)
Fluid overload (Metabolism and nutrition disorders) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 2 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (3)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0)
Autonomic nervous system imbalance (Nervous system disorders) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 2 (2)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Ageusia (Nervous system disorders) | 0 (0) | 1 (1)
Amnesia (Nervous system disorders) | 0 (0) | 1 (1)
Knee arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0)
Corona virus infection (Infections and infestations) | 0 (0) | 0 (0)
Extremity necrosis (Vascular disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-15): https://cdn.clinicaltrials.gov/large-docs/80/NCT02533180/Prot_001.pdf
  • Statistical Analysis Plan (2020-02-10): https://cdn.clinicaltrials.gov/large-docs/80/NCT02533180/SAP_000.pdf